CLINICAL TRIAL: NCT02784002
Title: A Phase II, Randomized, Open-Label, Active-Controlled Clinical Study to Investigate the Safety and Efficacy of SMT19969 (200mg BID) for 10 Days Compared With Fidaxomicin (200 mg BID) for 10 Days for the Treatment of Clostridium Difficile Infection (CDI)
Brief Title: A Study of Ridinilazole (SMT19969) Compared With Fidaxomicin for the Treatment of Clostridium Difficile Infection (CDI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Summit Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMT19969/C003
Record Dates: First submitted 2016-05-16; First posted 2016-05-26 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Clostridium Difficile Infection
MeSH Terms: conditions — Clostridium Infections | interventions — ridinilazole; Fidaxomicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ridinilazole (SMT19969) (Experimental): 200 mg capsule of Ridinilazole (SMT19969) twice a day for 10 days
  Interventions: Drug: Ridinilazole
- Fidaxomicin (Active Comparator): 200 mg tablet of Fidaxomicin twice a day for 10 days
  Interventions: Drug: Fidaxomicin

INTERVENTIONS:
Drug: Ridinilazole
  Other Names: SMT19969
  Arms: Ridinilazole (SMT19969)
Drug: Fidaxomicin
  Arms: Fidaxomicin

SUMMARY:
The purpose of this research study is to evaluate the safety and effectiveness of Ridinilazole (SMT19969) in treating C. difficile Infection (CDI).

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* Clinical diagnosis of CDI plus laboratory diagnostic test
* No more than 30 hours antimicrobial treatment for current CDI episode
* Female subjects of childbearing potential must use adequate contraception

Exclusion Criteria:

* Life-threatening or fulminant CDI
* Subjects with 2 or more episodes of CDI in the previous year
* Females who are pregnant or breastfeeding
* History of inflammatory bowel disease
* Co-administration of potent P-glycoprotein inhibitors
* Participation in other Clinical research studies within one month of screening
* Subjects that the Investigator feels are inappropriate for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (AEs) and serious adverse events (SAEs) to evaluate safety and tolerability | 30 days post End of Therapy

SECONDARY OUTCOMES:
To assess the pharmacokinetics of SMT19969 in patients with CDI by measuring the plasma, urine and fecal concentrations of SMT19969 | 12 days
To assess the qualitative and quantitative effect on the bowel flora of each subject using 16S ribosomal RNA sequencing, metagenomics and bioinformatic techniques | 40 days
Measure clinical cure rates at the Test of Cure (TOC) visit | 12 days
  Investigator assessed clinical response at the TOC visit (on day 12) with clinical cure defined as the resolution of diarrhoea (≤ 3 Unformed Bowel Movements (UBMs) per day) while on treatment that is maintained until the TOC visit.
Measure sustained clinical response (SCR) rates | 40 days
  SCR is defined as clinical cure at TOC and no recurrence of CDI within 30 days post end of treatment (EOT).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Summit Therapeutics
Locations (16):
- United States (5):
  - Laguna Hills, Laguna Hills, California
  - Ventura, Ventura, California
  - Idaho, Idaho Falls, Idaho
  - Butte, Butte, Montana
  - New Jersey, Somers Point, New Jersey
- Czechia (4):
  - Liberec, Liberec
  - Pardubice, Pardubice
  - Praha, Prague
  - Zlin, Zlín
- United Kingdom (7):
  - Leeds, Leeds
  - Liverpool, Liverpool
  - London, London
  - Manchester, Manchester
  - Newcastle Upon Tyne, Newcastle upon Tyne
  - Oxford, Oxford
  - Wigan, Wigan

IPD SHARING:
Plan to Share IPD: Undecided